CLINICAL TRIAL: NCT05099341
Title: DEPLIPIDO Study: Functional and Lipidomic Analysis of Plasma HDL in Patients With Depression Compared to Controls
Acronym: DepLIPIDO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHAUVET CRBFC-E 2019
Record Dates: First submitted 2021-10-04; First posted 2021-10-29 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients with recurrent depression with a number of depressive episodes ≥ 3 (Experimental)
  Interventions: Other: HDRS-17 depression scale; Biological: Blood sampling
- Patients with a first depressive episode (Experimental)
  Interventions: Other: HDRS-17 depression scale; Biological: Blood sampling
- Healthy, non-depressed subjects (Active Comparator)
  Interventions: Other: HDRS-17 depression scale; Biological: Blood sampling

INTERVENTIONS:
Other: HDRS-17 depression scale — Measuring the severity of depression
Biological: Blood sampling — 3 tubes of 5 ml

SUMMARY:
Depression is a disabling condition in terms of psychosocial alteration and also in terms of physical comorbidities. Depression doubles the risk of myocardial infarction compared with the general population, and this cardiovascular comorbidity leads to an increase in mortality in patients suffering from depression, even exceeding suicide-related mortality.

It is therefore important to better understand the mechanisms linking depression and cardiovascular disease.

Among the hypotheses that may account for the increased cardiovascular risk in patients with depression, lipid abnormalities are likely to play a crucial role.

Thus, qualitative and functional abnormalities in HDL lipoproteins are an important line of research, insofar as these lipid abnormalities have been recognized as important atherogenic abnormalities in populations at high cardiovascular risk, which is the case of patients with depression.

In this clinical, epidemiological and scientific context, a collaborative study undertaken by both the Department of Psychiatry of the Dijon Bourgogne University Hospital of and the INSERM LNC-UMR 1231 (PADYS) Laboratory of the UNIVERSITY OF BOURGOGNE FRANCHE-COMTE is an original translational research project, and the first study to perform a lipidomic analysis of HDL, coupled with a functional analysis of these lipoproteins in depression.

ELIGIBILITY:
Inclusion Criteria:

* FOR PATIENTS WITH RECURRENT DEPRESSION :

  * Patient who has provided oral consent
  * Adult with moderate to severe depression according to DSM-5 criteria (Hamilton HDRS-17 score ≥ 18), with a number of depressive episodes ≥ 3
* PATIENTS PRESENTING WITH A FIRST DEPRESSIVE EPISODE

  * Patient who has provided oral consent
  * Adult with moderate to severe characterized depression according to DSM-5 criteria (Hamilton HDRS-17 scale score ≥ 18) presenting with a first depressive episode.
* CONTROLS

  * Person who has provided oral consent
  * Adult who has never shown signs of depression

Exclusion Criteria:

* Person not affiliated with national health insurance
* Person subject to a measure of legal protection (curatorship, guardianship)
* Pregnant or breastfeeding women
* Adult unable to express consent
* Minors
* Person with a metabolic syndrome (according to NCEP/ATP-III criteria: 3 of the following 5 criteria: Waist circumference ≥ 102 cm in males and ≥ 88cm in females, Triglycerides > 1.50 g/L, HDL-Cholesterol < 0.40 g/L in H, HDL-Cholesterol < 0.50 g/L in F, Blood pressure ≥130/85mmHg, Fasting blood glucose ≥ 1.10 g/L),
* Person with type 1 or type 2 diabetes,
* Person with a mild depressive episode (HDRS-17<18),
* Person with concomitant antipsychotic treatment
* Person with bipolar disorder,
* Person with a moderate to severe alcohol use disorder according to DSM-5 criteria
* Person with schizophrenia,
* Person with a persistent delusional disorder,
* Person with an autism spectrum disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Measurement of cholesterol efflux by fluorescent method on THP-1 cell derived macrophages | At baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No